CLINICAL TRIAL: NCT00391027
Title: A Six Month, Open-Label Outpatient, Randomized Parallel Group Trial Assessing The Impact Of Dry Powder Inhaled Insulin (Exubera®) On Glycemic Control Compared To Insulin Glargine (Lantus®) In Patients With Type 2 Diabetes Mellitus Who Are Poorly Controlled On A Combination Of Two Or More Oral Agents
Brief Title: A Clinical Trial Comparing the Efficacy and Safety of Exubera® and Lantus®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171084
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Results first posted 2009-10-21 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes, insulin, glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin Glargine; Exubera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Glargine (Lantus®) (Active Comparator)
  Interventions: Drug: Insulin Glargine (Lantus®)
- Inhaled Human Insulin (Exubera®) (Active Comparator)
  Interventions: Drug: Inhaled Human Insulin (Exubera®)

INTERVENTIONS:
Drug: Insulin Glargine (Lantus®) — Patient will be randomized to Lantus® while remaining on pre-study oral hypoglycemic agents.
  Arms: Insulin Glargine (Lantus®)
Drug: Inhaled Human Insulin (Exubera®) — Patient will be randomized inhaled insulin while remaining on pre-study oral hypoglycemic agents.
  Arms: Inhaled Human Insulin (Exubera®)

SUMMARY:
To compare efficacy and safety of Exubera® vs Lantus® in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus, Type 2 on oral agents
* Age > 30 years

Exclusion Criteria:

* Severe Asthma, severe Chronic Obstructive Pulmonary Disease
* Smoking

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- Belgium (4):
  - Pfizer Investigational Site, Bornem
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Liège
- Finland (3):
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Lahti
  - Pfizer Investigational Site, Oulu
- France (6):
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Corbeil-Essonnes
  - Pfizer Investigational Site, La Rochelle
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Valenciennes
- Germany (8):
  - Pfizer Investigational Site, Altenburg
  - Pfizer Investigational Site, Eisenach
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hohenmölsen
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Neuss
  - Pfizer Investigational Site, Riesa
  - Pfizer Investigational Site, Wangen / Allgaeu
- Netherlands (5):
  - Pfizer Investigational Site, 's-Hertogenbosch
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, The Hague
  - Pfizer Investigational Site, Venlo
- Norway (5):
  - Pfizer Investigational Site, Hønefoss, Buskerud
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Jessheim
  - Pfizer Investigational Site, Lysaker
  - Pfizer Investigational Site, Skedsmokorset
- Poland (4):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Łask
- Spain (8):
  - Pfizer Investigational Site, A Coruña, A Coruña
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Huelva, Huelva
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Inca, Mallorca
  - Pfizer Investigational Site, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Pfizer Investigational Site, Alzira, Valencia
  - Pfizer Investigational Site, Valencia, Valencia
- Sweden (15):
  - Pfizer Investigational Site, Borås
  - Pfizer Investigational Site, Eksjö
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Härnösand
  - Pfizer Investigational Site, Helsingborg
  - Pfizer Investigational Site, Järfälla
  - Pfizer Investigational Site, Kristianstad
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Luleå
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Motala
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uddevalla
  - Pfizer Investigational Site, Umeå
  - Pfizer Investigational Site, Vaxjo
- Switzerland (2):
  - Pfizer Investigational Site, Bruderholz
  - Pfizer Investigational Site, Sankt Gallen

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171084&StudyName=A%20Clinical%20Trial%20Comparing%20the%20Efficacy%20and%20Safety%20of%20Exubera%AE%20and%20Lantus%AE

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of subjects randomized = 261; number of subjects treated (out of 261 randomized) = 257.
Groups:
- Inhaled Human Insulin (Exubera®): Pre-prandial inhaled insulin regimen administered three times a day (TID) using Exubera® Inhaler device; insulin packaged as 1 or 3 milligram (mg) dry powder insulin. Initial daily dose determined based on subject's body weight and divided into 3 doses administered prior to major meals. Pre-meal doses modified based on meal size and pre-prandial blood glucose readings. Subjects combined 1 and 3 mg doses before each meal to control post-prandial glycemia in addition to continuing their usual oral (PO) drugs at the pre-study doses unless clinical need justified a dose modification.
- Insulin Glargine (Lantus®): Insulin glargine (Lantus®) 10 International Units (IU) injected subcutaneously (SC) once daily (QD) at the same time of day (morning dose recommended) for the duration of the study (26 Weeks) using a pen device where available. Daily dose of insulin glargine modified based on glucose measurements at the discretion of the treating physician. Insulin glargine added initially to subject's usual oral regimen and was to be continued at pre-study doses unless clinical need justified a dose modification.
Period: Overall Study
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Started | 135 (Full Analysis Set = 134; 1 subject excluded; missing a baseline or postbaseline HbA1c measurement.) | 122 (Full Analysis Set = 121; 1 subject excluded; missing a baseline or postbaseline HbA1c measurement.)
Completed | 110 | 110
Not Completed | 25 | 12
Not completed — Adverse Event | 8 | 8
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 10 | 1
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®) | Total
Number analyzed (Participants) | 135 | 122 | 257
Age, Customized [Number; unit: participants]
  18 - 44 years | 8 | 3 | 11
  45 - 64 years | 78 | 71 | 149
  > = 65 years | 49 | 48 | 97
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 51 | 105
  Male | 81 | 71 | 152

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26
Description: Change (measured as percent): HbA1c at observation minus HbA1c at baseline. Primary objective to demonstrate non-inferiority of inhaled insulin compared to insulin glargine for glycemic control after 26 weeks of treatment not attainable due to early termination of study; analyses were descriptive and graphical.
Time Frame: Baseline, Week 26
Population: Full analysis set (FAS) all randomized subjects with at least 1 dose of study medication, baseline and post-baseline HbA1c measurement. Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 121
percent | -1.7 (1.19) | -1.4 (1.14)

2. Secondary Outcome: Change From Baseline in HbA1c Prior to Week 26
Description: Change (measured as percent) from baseline calculated as HbA1c at observation minus HbA1c at baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, and Week 18
Population: FAS; LOCF; (n) = number of subjects with analyzable data at observation for inhaled insulin and insulin glargine, respectively.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 121
percent
  Week 2 (n = 128, 108) | -0.4 (0.40) | -0.3 (0.40)
  Week 4 (n = 134, 121) | -0.8 (0.61) | -0.6 (0.58)
  Week 8 (n = 134, 121) | -1.3 (0.86) | -1.1 (0.85)
  Week 12 (n = 134, 121) | -1.6 (1.08) | -1.3 (0.99)
  Week 18 (n = 134, 121) | -1.7 (1.16) | -1.5 (1.11)

3. Secondary Outcome: Number of Subjects With HbA1c < 6.5 %
Description: Number of subjects with glycemic control HbA1c measurement of < 6.5 % at observation.
Time Frame: Week 26
Population: FAS
Measure: Number; unit: participants
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 121
participants | 37 | 23

4. Secondary Outcome: Number of Subjects With HbA1c < 7.0 %
Description: Number of subjects with glycemic control HbA1c measurement of < 7.0 % at observation.
Time Frame: Week 26
Population: FAS
Measure: Number; unit: participants
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 121
participants | 84 | 67

5. Secondary Outcome: Number of Subjects With HbA1c < 8.0 %
Description: Number of subjects with glycemic control HbA1c measurement of < 8.0 % at observation.
Time Frame: Week 26
Population: FAS
Measure: Number; unit: participants
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 121
participants | 121 | 108

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) Level
Description: FPG measured as milligrams/deciliter (mg/dl). Change from baseline calculated as FPG at observation minus FPG at baseline.
Time Frame: Baseline, Week 26
Population: FAS; LOCF.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 120
mg/dl | -30.6 (49.04) | -60.1 (51.95)

7. Secondary Outcome: Analysis of Home Blood Glucose Monitoring (HBGM) (7 & 8 Point)
Description: Blood glucose (BG) self-monitored by subject at home; measured at least once between Visits 2, 3 and between Visits 8, 9 (8-point: fasting, pre-meal, post-meal, bedtime, 2:00 am); between each visit: Visit 3 to 8 (7-point: fasting, post-meal, pre-lunch, pre-dinner, bedtime). Post-meal: 2-hour period after breakfast, lunch, dinner. Change: average overall absolute, pre-meal, and post-meal blood glucose = HBGM at observation minus HBGM at baseline; pre-meal to post-meal blood glucose = HBGM at post-meal minus HBGM at pre-meal.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 121
mg/dl
  Average overall absolute BG (n=101, 95) | -45.0 (46.26) | -43.7 (48.41)
  Average pre-meal BG (n=101, 95) | -38.1 (43.24) | -50.7 (47.54)
  Average post-meal BG (n=99, 91) | -64.5 (59.35) | -49.6 (58.33)
  Change from pre-meal to post-meal BG (n=99, 91) | -24.5 (35.28) | 1.6 (39.82)

8. Secondary Outcome: Number of Subjects With Hypoglycemic Events by Severity
Description: Number of subjects with hypoglycemic events by severity. Severe hypoglycemia: subject unable to treat self; exhibits a neurological symptom; and blood glucose <=2.72 mmol/L or blood glucose not measured but symptoms reversed with food intake, SC glucagon, or intravenous glucose. If all 3 criteria not met, hypoglycemia defined as mild or moderate.
Time Frame: Week 26
Population: FAS
Measure: Number; unit: participants
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 121
participants
  Week 26 Mild, Moderate | 26 | 32
  Week 26 Severe | 1 | 1

9. Secondary Outcome: Number of Events of Nocturnal Hypoglycemia
Description: Number of events of nocturnal hypoglycemia, incidence: midnight to 6:00 am. Hypoglycemia: characteristic symptoms of hypoglycemia with no blood glucose check; resolved with food intake, SC glucagon, or intravenous (IV) glucose; or symptoms with glucose <3.27 mmol/L (59 mg/dL); or any glucose measurement <=2.72 mmol/L (49 mg/dl). Severity of nocturnal glycemia not summarized.
Time Frame: Week 26
Population: FAS
Measure: Number; unit: events
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 121
events | 159 | 81

10. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline calculated as body weight at observation minus body weight at baseline.
Time Frame: Baseline, Week 26
Population: FAS; LOCF.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 125 | 118
kilograms (kg) | 2.2 (3.57) | 1.1 (3.43)

11. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: BMI measured as kilograms per meter squared (kg/m2). Change calculated as BMI at observation minus BMI at baseline.
Time Frame: Baseline, Week 26
Population: FAS; LOCF.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 125 | 118
kg/m2 | 0.7 (1.24) | 0.4 (1.20)

12. Secondary Outcome: Number of Subjects Discontinued Due to Insufficient Clinical Response
Description: Number of subjects discontinued due to signs and symptoms of persistent hyperglycemia or HbA1c > 12.0 % or frequent and unexplained severe hypoglycemic events (> 3 events per month for 2 or more months); subject's HbA1c not < = 7 % at Week 12.
Time Frame: Week 26
Population: Safety population: all subjects who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 135 | 122
participants | 3 | 0

13. Secondary Outcome: Change From Baseline in Treatment Satisfaction, Quality of Life, and Mental Health
Description: Subject reported outcomes for Diabetes Treatment Satisfaction Questionnaire-Status (DTSQs), DTSQ-change, Patient Satisfaction with Insulin Therapy-16 item, Mental Health Inventory-17 item, and Euro Quality of life 5-Dimensions (EuroQol 5-D) Questionnaire not summarized due to cancellation of Exubera® program.
Time Frame: Week 26
Reporting Status: Not Posted

14. Secondary Outcome: Continuous Glucose Monitoring System (CGMS) 24-hour Glucose Profile in a Subset of Patients
Description: The mean of the 24-hour mean and the mean of the 24-hour standard deviation (SD) (variability around the average glucose concentration) calculated on glucose values (mg/dl) collected during inpatient evaluation of glycemic stability. Interstitial glucose assessed at 5 minute intervals starting pre-supper on Day 1 of evaluation; ending on Day 3 pre-breakfast. Analysis is on data generated between 6:00 am on Day 2 and 6:00 am on Day 3.
Time Frame: Baseline, Week 26
Population: FAS; (n) = number of subjects with analyzable data at observation for inhaled insulin and insulin glargine, respectively. Revised table rectifies a programming code error that was determined post-Clinical study report (CSR) approval.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 134 | 121
mg/dl
  Week 26: 24-hour mean (n=14, 12) | 107.6 (18.46) | 102.1 (18.02)
  Week 26: 24-hour SD (n=14, 12) | 33.7 (17.22) | 30.7 (8.09)

15. Secondary Outcome: Change From Baseline in Cardiovascular (CV) Biomarkers - High Sensitive C-reactive Protein (Hs-CRP)
Description: Change from baseline in CV biomarker hs-CRP (milligrams per deciliter [mg/dl]) calculated as hs-CRP at observation minus hs-CRP at baseline.
Time Frame: Baseline, Week 26
Population: FAS; LOCF.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 106 | 98
mg/dl | 0.2 (1.92) | -0.1 (1.56)

16. Secondary Outcome: Change From Baseline in CV Biomarkers - Interleukin 6 (IL-6)
Description: Change from baseline in IL-6 (picograms per milliliter [pg/ml]) calculated as IL-6 at observation minus IL-6 at baseline.
Time Frame: Baseline, Week 26
Population: FAS; LOCF.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 55 | 61
pg/ml | -1.1 (4.05) | -2.4 (10.41)

17. Secondary Outcome: Change From Baseline in CV Biomarkers - Thrombin-antithrombin Complexes (Tat-complexes)
Description: Change from baseline in tat-complexes (nanograms per milliliter [ng/ml]) calculated as tat-complexes at observation minus tat-complexes at baseline.
Time Frame: Baseline, Week 26
Population: FAS; LOCF.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 31 | 18
ng/ml | -3.4 (10.00) | -40.4 (166.90)

18. Secondary Outcome: Change From Baseline in CV Biomarkers - Soluble Tissue Factor (STF)
Description: Change from baseline in soluble tissue factor (pg/ml) calculated as STF at observation minus STF at baseline.
Time Frame: Baseline, Week 26
Population: FAS; LOCF.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Number analyzed (Participants) | 2 | 5
pg/ml | 230.2 (279.92) | 170.4 (174.07)

19. Secondary Outcome: Change From Baseline in Urinary Free 8-iso Prostaglandin F2-alpha (α) in a Subset of Subjects
Description: Urinary free 8-iso prostaglandin F2-alpha (α): compare glucose fluctuations and activation of oxidative stress as assessed by urinary isoprostanes in a subset of subjects randomized to either Exubera® or subcutaneous insulin glargine. The substudy was offered to all subjects. Data not summarized due to cancellation of Exubera® program.
Time Frame: Baseline, Week 26
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Inhaled Human Insulin (Exubera®) | Insulin Glargine (Lantus®)
Serious Adverse Events (participants affected / at risk) | 8/135 | 10/122
Other Adverse Events (participants affected / at risk) | 105/135 | 81/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Human Insulin (Exubera®) (N=135) | Insulin Glargine (Lantus®) (N=122)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Myotonia (Nervous system disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Human Insulin (Exubera®) (N=135) | Insulin Glargine (Lantus®) (N=122)
Angina pectoris (Cardiac disorders) | 1 | 2
Vision blurred (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Chest pain (General disorders) | 2 | 0
Fatigue (General disorders) | 5 | 4
Oedema (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 9 | 2
Bronchitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 18 | 20
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Weight increased (Investigations) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 95 | 65
Increased appetite (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 7 | 3
Paraesthesia (Nervous system disorders) | 3 | 0
Sciatica (Nervous system disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Hypertension (Vascular disorders) | 6 | 2

LIMITATIONS AND CAVEATS:
Enrollment period concluded earlier than planned due to cancellation of Exubera® program by sponsor; enrollment was undersized to meet requirements of its inferential objectives. Revised analysis approach was descriptive with no inferential analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.